CLINICAL TRIAL: NCT02254902
Title: Physical Activity and Education to Reduce Cancer Risk Among Somali Women (Ladnaan Project)
Brief Title: Physical Activity and Education Program for Somali Women
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Changes in funding status
Sponsor: University of California, San Diego (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Kate Murray, PhD, MPH, Assistant Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACS-MRSG-13-069
Record Dates: First submitted 2014-09-29; First posted 2014-10-02 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Sedentary Lifestyle
Keywords: sedentary lifestyle; physical activity; Somali women; prevention
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical Activity (Experimental): Participants in the Physical Activity intervention arm of the study receive culturally-modified, materials through participation in 12 weekly 1-.5-hour sessions focused on increasing daily step counts and bouts of moderate intensity physical activity. The group sessions include participation in different forms of physical activity as well as group discussions on the barriers and opportunities for increasing physical activity in daily life.
  Interventions: Behavioral: Physical Activity intervention
- Wait List Control (No Intervention): Participants in the Wait List Control will be offered the program after a 3-month wait period. While waiting for the program, participants are offered to attend monthly sessions on various wellness and prevention topics.

INTERVENTIONS:
Behavioral: Physical Activity intervention — The Physical Activity intervention is a 3-month group-based program based on an efficacious physical activity intervention that has been culturally adapted for use with adult Somali women. The program targets increased physical activity through educational and experiential opportunities.
  Arms: Physical Activity

SUMMARY:
There is a significant need for culturally adapted and effective health education programs to address rising rates of obesity and chronic disease concerns for refugee communities. Physical activity has been identified as an important prevention tool to prevent numerous chronic health conditions. This research tests the feasibility and acceptability of a culturally adapted physical activity intervention for sedentary adult Somali women. Study participants will be randomized to a 3-month physical activity program or a wait-list control group. The primary outcome is increases in physical activity between baseline and the end of the program as measured by pedometer.

DETAILED DESCRIPTION:
Participants in the physical activity program will participate in 12 weekly 1.5-hour sessions focused on increasing physical activity. The group sessions will include participating in physical activity as well as group discussions on the barriers and opportunities for increasing physical activity in their daily life. The 12-week program covers educational topics related to physical activity (e.g. overcoming barriers to activity, exercising safely, relapse prevention strategies) and the program gradually increases the amount of physical activity completed during the group sessions over the course of the 12 weeks. Over a 3-month wait period, individuals in the wait-list control group will be offered monthly sessions on health and wellness topics before being offered the physical activity program. Measurement visits will occur at baseline, at the end of the12-week program, and approximately 12-weeks after the end of the intervention. During the measurement sessions participants will complete assessments related to their physical activity and other health behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary (less than 90 minutes per week of moderate or vigorous physical activity)
* Self-identify as Somali
* Planning on living in the area for the next 6 months
* Ability to attend 12-weeks of in-person group sessions at a designated community site

Exclusion Criteria:

* Currently pregnant or within 3 months of delivery
* BMI greater than or equal to 40
* Medical conditions or physical problems that interfere with physical activity or require medical supervision to exercise
* Have another member of the household participating in the study
* Employment by one of the collaborating organizations

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in physical activity as measured by pedometer from baseline to 3 months | Baseline and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kate E Murray, PhD, MPH, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, La Jolla, California, United States